CLINICAL TRIAL: NCT03995992
Title: Evaluation of the Impact of Diving Training on Recovery in a Cohort of Veterans Suffering of PTSD: an Exploratory Clinical Control Trial
Brief Title: Benefits of Diving Training on Recovery for Veterans Suffering of Chronic PTSD: an Exploratory Study
Acronym: cognidive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Recherche Biomedicale des Armees (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRBA
Record Dates: First submitted 2019-05-18; First posted 2019-06-24 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Stress Disorder, Combat
MeSH Terms: conditions — Combat Disorders

STUDY DESIGN:
Intervention Model Description: two groups whih differ by the type of sport training: multisport versus diving
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multi sport (Active Comparator): During 10 days, each morning, from 9 am to 12 pm, participants had sporting activities: mountain walking, mountain biking, climbing, canyoning and collective orienteering running. From 3 pm, they had individual and collective practical workshops based on PTSD psychoeducation, human resources competences and coaching, including a curriculum vitae workshop. During their free time, they could take part in collective activities like table football, pool, party games or have a rest. Relaxation exercises were proposed every day after the sporting activity and before dinner.
  Interventions: Behavioral: sport
- diving (Experimental): During 10 days, each morning, from 9 am to 12 pm, participants had diving activities. From 3 pm, they had individual and collective practical workshops based on PTSD psychoeducation, human resources competences and coaching, including a curriculum vitae workshop. During their free time, they could take part in collective activities like table football, pool, party games or have a rest. Relaxation exercises were proposed every day after the sporting activity and before dinner.
  Interventions: Behavioral: sport

INTERVENTIONS:
Behavioral: sport — 10 days of sport (diving or multisport), once training per day

SUMMARY:
Patients suffering from Chronic Posttraumatic Stress Disorder (PTSD) have difficulties in executive cognition that hinder their quality of life and make it difficult to recovery and to reintegrate them socially and professionally. These difficulties are particularly important for soldiers suffering from chronic PTSD.

The literature suggests that diving may be a complementary approach to improving cognition, in addition to its benefits on the quality of life of patients with chronic PTSD. It appears to be an intervention of interest to improve the successful recovery for veterans with PTSD compared to a multi-sport practice.

DETAILED DESCRIPTION:
A French military rehabilitation program proposes the broadening of the relationships between recovery and reintegration by incorporating approaches in the field of positive psychology for soldiers with chronic PTSD. This program was organized for a group of 10 veterans for 10 days. Each morning, from 9 am to 12 pm, participants had sporting activities: mountain walking, mountain biking, climbing, canyoning and collective orienteering running. From 3 pm, they had individual and collective practical workshops based on PTSD psychoeducation, human resources competences and coaching, including a curriculum vitae workshop.

The investigators aims to compare this program included multisport practice with the same praogram included diving instead of multi-sport to evaluate the impact to recovery at one year

ELIGIBILITY:
Inclusion Criteria:

* veterans
* having a chronic PTSD evaluated by a psychiatrist All soldiers included in this study were on sick leave for at least 6 months due to chronic PTSD and were waiting for a military invalidity committee pension. They were all engaged in the first step of the Omega project and had a nine-day HRT training session planned

Exclusion Criteria:

* the psychiatrist did not consider the clinical state appropriate enough to take part in the omega project

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-08 (Actual); Primary Completion 2022-11-28 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
status of professional reinsertion (having a job or not) | one year after the intervention (sport training)
  Rate of professional reinsertion

SECONDARY OUTCOMES:
PTSD symptoms | two times points ; change were assessed between before and after the sport training (eg. before and 10 days after)
  self-report scale: the post-traumatic checklist 5 (PCL5) threshold=33
cognitive symptoms | two times points ; change were assessed between before and after the sport training (eg. before and 10 days after)
  self report scale: the Montreal Cognive Assessment (MOCA) threshold=27

OTHER OUTCOMES:
inflammatory level | two times points ; change were assessed between before and after the sport training (eg. before and 10 days after)
  salivary cytokines

CONTACTS AND LOCATIONS:
Overall Officials: marion trousselard, Principal Investigator — Institut de Recherche Biomedicale des Armees
Locations (2):
- France (2):
  - Marion, Brétigny-sur-Orge, Not in US/Canada
  - anne-sophie Pellen, Paris, Not in US/Canada

IPD SHARING:
Plan to Share IPD: No